CLINICAL TRIAL: NCT06536803
Title: Effects of High Load Strength Training With and Without Tissue Specific Planter Facia Stretching Exercise on Pain Range of Motion and Functional Disability Among the Athletes With Planter Fasciitis
Brief Title: Effects of High Load Strength Training With and Without Tissue Specific Planter Facia Stretching With Planter Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0471
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Plantar Fascitis; Resistance Training; Muscle Stretching Exercises
Keywords: plantar heel pain,High-load strength training,

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial
Who Masked: Outcomes Assessor
Masking Description: single outcome assessor who will take the reading is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-load strength training with tisssue specific plantar fascia stretching exercise (Active Comparator): Experimental group will receive high load strength training and Tissue-specific plantar fascia stretching exercise and routine physiotherapy. Pain, range of motion and functional disability will be measured before session, immediate effect after first session,then after 06 weeks (18 session) with high load strength training maximum repetition 12 RM with 3 sets in alternative days in each set minimum 2 mint rest interval and tissue specific plantar fascia stretching exercise perform for 10 times for 10 sec, after 12 weeks (36 sessions) with high load strength training maximum repetition 10 RM with 4 sets in alternative days in each set minimum 2 mint rest interval tissue specific plantar fascia stretching exercise perform for 10times
  Interventions: Other: high load strength training and Tissue-specific plantar fascia stretching exercise for 12 weeks
- high-load strength training with routine physiotherapy (Active Comparator): active compator group will then receive high load strength training and routine physiotherapy ultrasonic therapy
  Interventions: Other: high-load strength training with routine physiotherapy

INTERVENTIONS:
Other: high load strength training and Tissue-specific plantar fascia stretching exercise for 12 weeks — high load strength training and Tissue-specific plantar fascia stretching exercise for 12 weeks
  Arms: high-load strength training with tisssue specific plantar fascia stretching exercise
Other: high-load strength training with routine physiotherapy — high load strength training with routine physiotherapy for 12 weeks
  Arms: high-load strength training with routine physiotherapy

SUMMARY:
The rationale behind examining the synergistic impacts of high load strength training and tissues pecific plantar fascia stretching activities in athletes diagnosed with plantar fasciitis arises from an acknowledged deficiency in the existing body of scholarly research.Study design will be Randomized Control Trial. The study will be completed in 10 months after Synopsis Approval.The study will be carried in sports clubs of MOTH Mirpur AJK. Convenient Sampling will be used. Data Collection Tools will be used named as VAS, Functional foot index (FFI), and Goniometry used for Pain, functional disability and range of motion will be measured respectively before and after the intervention

DETAILED DESCRIPTION:
Population is divided into 2 groups: Group A and Group B. Both groups will be given a patient evaluation sheet and thickness of planter fascia will be already measured by Ultrasound. Group A will then receive high load strength training and routine physiotherapy. Group B will receive high load strength training and Tissue-specific plantar fascia stretching exercise and routine physiotherapy. Pain, range of motion and functional disability will be measured before session, immediate effect after first session, then after 06 weeks (18 session) with high load strength training maximum repetition 12 RM with 3 sets in alternative days in each set minimum 2 mint rest interval and tissue specific plantar fascia stretching exercise perform for 10 times for 10 sec, after 12 weeks (36 sessions) with high load strength training maximum repetition 10 RM with 4 sets in alternative days in each set minimum 2 mint rest interval tissue specific plantar fascia stretching exercise perform for 10 times for 10 sedate will be entered and analyzed by SPSS version 21. Statistical significance will be p=0.05 Descriptive statistics: Frequency tables, pie charts, bar charts will be used.

ELIGIBILITY:
Inclusion Criteria:

* Only Male Athletes
* Prediagnosed Patients suffering from Plantar fasciitis referred from Orthopedic.
* History of inferior heel pain atleast 2 weeks before enrollement.
* Pain on palpation of Medial calcaneal Tubercle/proximal Plantar Fascia.
* All participants with in the age group between 20-35 yrs.
* Patients who are willing to particiapate in the study.
* Heel pain syndrome

Exclusion Criteria:

* History of any systemic disease
* Heel and skin infection
* History of prior Surgery
* Corticosteroid injection for Plantar fasciitis within previous 06 momths;
* Any known malignancy /neoplasma involved side.
* Diagnosed/known psychiatric illness

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-09-26 (Estimated)

PRIMARY OUTCOMES:
Range of motion | 0 week,6 weeks ,12 week
  will be measured through goniometer
functional disability measured through Foot Function Index | 0 week,6 weeks ,12 week
  will be measured through Foot Function Index

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad ilyas, Principal Investigator — Riphah International University
Locations (1):
- Youth foot ball club,MOTH, Mirpur Mathelo, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID 21916393
- [Background] Rathleff MS, Molgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports. 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID 25145882
- [Background] Huffer D, Hing W, Newton R, Clair M. Strength training for plantar fasciitis and the intrinsic foot musculature: A systematic review. Phys Ther Sport. 2017 Mar;24:44-52. doi: 10.1016/j.ptsp.2016.08.008. Epub 2016 Aug 18. PMID 27692740
- [Background] Digiovanni BF, Nawoczenski DA, Malay DP, Graci PA, Williams TT, Wilding GE, Baumhauer JF. Plantar fascia-specific stretching exercise improves outcomes in patients with chronic plantar fasciitis. A prospective clinical trial with two-year follow-up. J Bone Joint Surg Am. 2006 Aug;88(8):1775-81. doi: 10.2106/JBJS.E.01281. PMID 16882901
- [Background] Rompe JD, Furia J, Cacchio A, Schmitz C, Maffulli N. Radial shock wave treatment alone is less efficient than radial shock wave treatment combined with tissue-specific plantar fascia-stretching in patients with chronic plantar heel pain. Int J Surg. 2015 Dec;24(Pt B):135-42. doi: 10.1016/j.ijsu.2015.04.082. Epub 2015 May 1. PMID 25940060
- [Background] Neufeld SK, Cerrato R. Plantar fasciitis: evaluation and treatment. J Am Acad Orthop Surg. 2008 Jun;16(6):338-46. doi: 10.5435/00124635-200806000-00006. PMID 18524985